CLINICAL TRIAL: NCT00123383
Title: Randomised Placebo-Controlled Trial of Modafinil for Cocaine Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); Kirketon Road Centre, Sydney Hospital (Unknown); St Vincent's Hospital, Sydney (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HREC05023
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2006-07

CONDITIONS: Cocaine Dependence
Keywords: Modafinil; Cocaine Dependence; Randomised placebo-controlled trial
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The study aims to evaluate the safety and efficacy of modafinil (200 mg/day) over 10 weeks plus a tailored cognitive behavioural therapy program in the treatment of cocaine dependence.

DETAILED DESCRIPTION:
Modafinil is a novel wake promoting agent approved in Australia for the treatment of narcolepsy. Preliminary studies have suggested that modafinil may have value in the treatment of psychostimulant dependence through positive effects on mood, sleep patterns, concentration, fatigue and drug craving. It appears to be well tolerated with a low abuse liability. Thirty dependent cocaine users will be randomised to 2 equal groups. The experimental group will receive modafinil 200 mg/day for 10 weeks and a tailored cognitive behavioural therapy program. The control group will receive placebo under equivalent conditions. Primary outcome will be a between group comparison of cocaine negative urine samples collected over the 10 week study period. Adverse events, side effects, compliance, retention, self reported health, psychosocial and drug use outcomes will also be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV cocaine dependence diagnosis
* Cocaine positive urine sample at intake
* Regular current cocaine use (2-3 days per week)
* Aged 18 years or older

Exclusion Criteria:

* Pregnant or nursing females
* Concurrent uncontrolled physical or mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-07; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Urinalysis negative for cocaine over 10 weeks | 10 weeks
Adverse events | 10 weeks
Compliance | 10 weeks
Retention | 10 weeks

SECONDARY OUTCOMES:
Self reported drug use | 10 weeks
Health outcomes | 10 weeks
Psychosocial outcomes | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Mattick, PhD, Principal Investigator — University of New South Wales
Locations (2):
- Australia (2):
  - Alcohol & Drug Services, St Vincent's Hospital, Darlinghurst, New South Wales
  - Kirketon Road Centre, Sydney Hospital, Darlinghurst, New South Wales

REFERENCES:
- [Derived] Shearer J, Shanahan M, Darke S, Rodgers C, van Beek I, McKetin R, Mattick RP. A cost-effectiveness analysis of modafinil therapy for psychostimulant dependence. Drug Alcohol Rev. 2010 May;29(3):235-42. doi: 10.1111/j.1465-3362.2009.00148.x. PMID 20565514